CLINICAL TRIAL: NCT05698225
Title: Characterising Pneumococcal Carriage and Immunity in People Living With HIV in Blantyre, Malawi, Following Experimental Pneumococcal Inoculation
Brief Title: Experimental Pneumococcal Carriage in People Living With HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EHPC in PLHIV
Record Dates: First submitted 2022-11-14; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-11

CONDITIONS: Pneumococcus; Pneumonia; Hiv
MeSH Terms: conditions — Pneumonia; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inoculation with Streptococcus pneumoniae serotype 6B (Experimental): Participants will be inoculation with a controlled concentration of full sequenced, fully antibiotic sensitive Streptococcus pneumonia serotype 6B
  Interventions: Other: Streptococcus pneumoniae serotype 6B

INTERVENTIONS:
Other: Streptococcus pneumoniae serotype 6B — A controlled concentration of streptococcus pneumoniae serotype 6B is placed in both nares of participants

SUMMARY:
The goal of this experimental pneumococcal carriage study is to to characterise rates and determinants of experimental pneumococcal carriage in PLHIV.

The main questions it aims to answer are:

* can PLHIV be experimentally inoculated with pneumococcus in a safe manner?
* what are the immunological determinants of pneumococcal carriage in PLHIV compared to HIV-negative participants?
* how do the pneumococcal carriage dynamics differ between PLHIV and HIV-negative participants?

Participants will be inoculated intranasally with a controlled concentration of pneumococcus after which they will be monitored for 21 days during which nasal and systemic immune dynamics and pneumococcal carriage dynamics will be evaluated. At the end of the study any participants exhibiting carriage will have the pneumococcus cleared with antibiotics.

DETAILED DESCRIPTION:
The EHPC has been established at the Malawi-Liverpool Wellcome centre (MLW) and demonstrated acceptability and feasibility in this setting. To date, over 250 participants have been enrolled on the EHPC at MLW without any study complications. Participants will be inoculated in both nostrils with a controlled concentration of penicillin-sensitive Streptococcus pneumoniae. Participants will be followed up for 25 days following inoculation during which sampling will occur at established time-points to establish pneumococcal carriage and immune cell/immunoglobulin dynamics. After 21 days, participants who demonstrate pneumococcal carriage will commence an antibiotic course to clear the bacteria (participants may be advised by the clinical study team to commence antibiotics earlier if they develop any symptoms of pneumococcal disease). Participants will remain under close observation in study accommodation for the first 3 days following inoculation, and will then be monitored daily at home via text message and telephone calls. A final health-check and exit interview will be conducted on day 25 to evaluate participant satisfaction with study participation. The overall objective is to characterise rates and determinants of experimental pneumococcal carriage in PLHIV in Blantyre, Malawi in order to inform vaccine evaluations and vaccine policy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 to 45 years old
* Fluent spoken and written Chichewa or English
* Able to give informed written consent
* Access to a functional mobile phone
* Establish on antiretroviral therapy for ≥2 years (if PLHIV)
* Viral load below the lower limit of detection (<LDL) at screening (if PLHIV)
* CD4 count over 350 cells/mm³ at screening (if PLHIV)

Exclusion Criteria:

* HIV-associated hospitalisation and/or treatment for major illness in preceding 2 years
* Currently under investigation for HIV-associated weight-loss, chronic diarrhoea, chronic cough, or another unexplained symptom
* Previous illness caused by pneumococcus
* Additional condition or medication impairing immune response or increasing risk of pneumococcal disease
* Living in close contact with an individual vulnerable to pneumococcal disease
* Allergy to penicillin
* Acute illness in 7 days preceding inoculation
* Antibiotic course in last 2 weeks (excluding prophylactic co-trimoxazole in PLHIV)
* Pregnant or trying to conceive
* Involved in another clinical study (unless observational or in follow-up)
* Current regular cigarette smoking (5+ cigarettes per week)
* Natural carrier of pneumococcus serotype 6B at screening visit
* Participants without a guardian

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with pneumococcal carriage in the nasopharynx post-inoculation | From inoculation up to 21 days post-inoculation
  Measured by classic culture and PCR-based methods

SECONDARY OUTCOMES:
Average pneumococcal carriage density in the nasopharynx post-inoculation | From inoculation up to 21 days post-inoculation
  Measured by classic culture and PCR-based methods
Nasal immunoglobulin concentration at baseline | Baseline
  Measured in nasal fluid
Change in nasal immunoglobulin concentration following inoculation | Baseline to 21 days post-inoculation
  Measured in nasal fluid
Density of immune cells in the nasal mucosa at baseline | Baseline
  Immune cell to epithelial cell ratio measured in nasal mucosal cell samples
Change in density of immune cells in the nasal mucosa following inoculation | Baseline up to 21 days post-inoculation
  Immune cell to epithelial cell ratio measured in nasal mucosal cell samples
Immune cell activation activation in the nasal mucosa at baseline | Baseline
  Concentration of markers of immune cell activation measured in nasal fluid and cell samples
Change in immune cell activation in the nasal mucosa following inoculation | Baseline up to 21 days post-inoculation
  Concentration of markers of immune cell activation measured in nasal fluid and cell samples

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gordon, MA MD, Principal Investigator — Malawi-Liverpool Wellcome Centre
Locations (1):
- Malawi-Liverpool Wellcome City, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No